CLINICAL TRIAL: NCT04325451
Title: An Observational Study to Determine Lifestyle, Biophysical and Environmental Risk Factors in the Development of Early-onset Pediatric Atopic Dermatitis
Brief Title: Comprehending Atopic Risk Elements
Acronym: CARE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: MYOR Ltd. (Industry)
Collaborators: Meir Medical Center (Other); The Baruch Padeh Medical Center, Poriya (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0244-19-MMC
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Skin barrier impairment and familial atopy have been implicated as crucial risk factors for the development of atopic dermatitis (AD). Additional risk factors have been explored, including gestational weight, height, age, familial smoking habits, proximity to urban centers and others. However, a comprehensive study focusing on the entire spectrum of risk factors has yet to be undertaken. Such a study could enable predictive capabilities able to inform medical professionals as to a newborn's inherent risk to develop AD, and potentially recommend appropriate preventative modalities to prevent or delay disease onset.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy newborn delivered in a hospital setting more than 24 hours prior to enrollment & less than 120 hours prior to enrollment
2. Term and near term newborns born between 34+0 and 42+0 weeks gestational age
3. Mothers must be aged >18 years
4. Parents' ability to complete questionnaire(s) at defined times throughout study duration
5. Parents or legal guardian provide informed written consent

Exclusion Criteria:

1. Preterm birth prior to 34+0 weeks gestation
2. Less than 12 hours out of the incubator
3. Neonate has undergone major surgery or intends to undergo major surgery in the coming 14 days
4. Neonate has an existing widespread skin condition that would make the detection and/or assessment of eczema difficult
5. Neonate has been administered oral or parenteral antibiotics from birth until study enrollment
6. Neonate has a serious health issue which, at parent or investigator discretion, would make it difficult for the neonate or parents to take part in the trial
7. Any other reason that, in the opinion of the investigator, prevents the subject from participating in the study or compromise the patient safety

Ages: 24 Hours to 120 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonates will be recruited from maternity wards amongst the general population within the first five days of life
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
To determine whether MyOR's Precision Infant Care (PIC) Algorithm accurately predicts the risk of developing atopic dermatitis | 24 months
  Evaluated using MyOR's Precision Infant Care (PIC) Algorithm V1.0

SECONDARY OUTCOMES:
To determine whether the combined information of familial history of atopy, TEWL, and other risk factors can effectively predict the risk of developing AD at six months of age. | 6 months
  Evaluated using the UK refinement of the Hanifin and Rajka diagnostic criteria for atopic eczema.
To determine whether the combined information of familial history of atopy, TEWL, and other risk factors can effectively predict the risk of developing AD at two years of age. | 24 months
  Evaluated using the UK refinement of the Hanifin and Rajka diagnostic criteria for atopic eczema.
To determine whether the combined information of familial history of atopy, TEWL, and other risk factors can effectively predict the severity of AD | 6 months
  Assessed using the Patient-Oriented Eczema Measure (POEM) questionnaire and accompanying scoring criteria.
To determine whether the combined information of familial history of atopy, TEWL, and other risk factors can effectively predict the severity of AD | 12 months
  Assessed using the Patient-Oriented Eczema Measure (POEM) questionnaire and accompanying scoring criteria.
To determine whether the combined information of familial history of atopy, TEWL, and other risk factors can effectively predict the severity of AD | 24 months
  Assessed using the Patient-Oriented Eczema Measure (POEM) questionnaire and accompanying scoring criteria.
3. To determine whether the combined information of familial history of atopy, TEWL, and other risk factors can effectively predict the age of onset of AD | 24 months
  Evaluated using the UK refinement of the Hanifin and Rajka diagnostic criteria for atopic eczema.
To determine whether the combined information of familial history of atopy, TEWL, and other risk factors can effectively predict the risk of developing food allergies | 12 months
  Evaluated using the 2010 U.S. Food and Drug Administration Food Safety Survey Questionnaire
To determine whether the combined information of familial history of atopy, TEWL, and other risk factors can effectively predict the risk of developing food allergies | 24 months
  Evaluated using the 2010 U.S. Food and Drug Administration Food Safety Survey Questionnaire
To determine whether MyOR's Precision Infant Care (PIC) Algorithm accurately predicts the risk of developing atopic dermatitis | 12 months
  Evaluated using MyOR's Precision Infant Care (PIC) Algorithm V1.0
To determine whether MyOR's Precision Infant Care (PIC) Algorithm accurately predicts the risk of developing food allergies | 24 months
  Evaluated using MyOR's Precision Infant Care (PIC) Algorithm V1.0
To determine whether the combined information of familial history of atopy, TEWL, and other risk factors can effectively predict the risk of development AD at one year of age | 12 months
  Evaluated using the UK refinement of the Hanifin and Rajka diagnostic criteria for atopic eczema. .

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Smolkin, MD, Principal Investigator — Poriah Medical Center; Tzofia Bauer, MD, Principal Investigator — Meir Medical Center
Locations (2):
- Israel (2):
  - Meir Medical Center, Kfar Saba
  - Poriya Medical Center, Tiberias

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brandwein M, Gamrasni K, Landau T, Bauer-Rusek S, Smolkin T. Nurture, not nature: Impaired skin barrier in infants born to urban households. Pediatr Allergy Immunol. 2022 Oct;33(10):e13868. doi: 10.1111/pai.13868. No abstract available. PMID 36282128